CLINICAL TRIAL: NCT03171688
Title: Risk Factors for Nausea and Vomiting After Cesarean: Observational Prospective Study
Brief Title: Risk Factors for Nausea and Vomiting After Cesarean
Status: Completed | Type: Observational
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, Head of Anesthesiology, Brasilia University Hospital
Other Study IDs: NVPOCesarianasGabriel2017
Record Dates: First submitted 2017-05-27; First posted 2017-05-31 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative Nausea and Vomiting; cesarean; risk factors
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modeling: It is the cohort that will be used for selecting risk factors and models for predicting postoperative nausea and vomiting.
- Validation: It is the cohort that will be used for validation of risk factors and models selected in the modeling group.

SUMMARY:
Investigators will observe the incidence of post-cesarean nausea or vomiting and try to associate it with some risk factors.

DETAILED DESCRIPTION:
A single prospective cohort of women submitted to cesarean section who received spinal anesthesia will be assessed for the proposed risk factors and the incidence of nausea or vomiting will be observed during the first 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean section indicated
* Spinal anesthesia indicated

Exclusion Criteria:

* Cesarean section did not occur
* Spinal anesthesia was not provided
* Another spinal technique was added to spinal

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women with indication for cesarean section in the University Hospital of University of Brasilia.
Sampling Method: Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Nausea or vomiting | 48 hours.
  The occurrence of postoperative nausea or vomiting, reported by the patient or witnessed by a healthcare provider during the first 48 hours after the cesarean. It is a dichotomic (true or false) outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel MN Guimaraes, MD, Study Chair — University of Brasilia
Locations (1):
- University Hospital of Brasilia University, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Plan to share excel sheets to allow meta-analysis.

DOCUMENTS (2):
  • Study Protocol (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03171688/Prot_000.pdf
  • Informed Consent Form (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03171688/ICF_001.pdf